CLINICAL TRIAL: NCT02740361
Title: International Deprexis Trial in Multiple Sclerosis (IDEMS) - a Multicenter Randomized Controlled Trial
Brief Title: Online Program to Reduce Depression in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: National Multiple Sclerosis Society (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Cedars-Sinai Medical Center (Other); University of Missouri, Kansas City (Other); Penn State University (Other); King's College London (Other); University Medical Center Goettingen (Other); NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Friedemann Paul, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDEMS; RG-1507-05418 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2016-04-12; First posted 2016-04-15 (Estimated); Last update posted 2025-05-20 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Deprexis (Experimental): This group will receive access to the web-based Deprexis program, an online tool based on principles of cognitive behavioral therapy. Contents include (1) psychoeducation, (2) behavioral activation, (3) cognitive modification, (4) mindfulness and acceptance, (5) interpersonal skills, (6) relaxation, physical exercise and lifestyle modification, (7) problem solving, (8) expressive writing and forgiveness, (9) positive psychology, and (10) emotion-focused interventions.
  Interventions: Behavioral: Deprexis, DeprexisPlus
- DeprexisPlus (Experimental): This group will receive the web-based Deprexis program (see above) plus scheduled e-mail contact (1x/week)
  Interventions: Behavioral: Deprexis, DeprexisPlus
- Waitlist Control (No Intervention): Participants randomized to the control group will wait for access to the Deprexis program (waitlist control) for 6 months. After the 6-month waiting period, participants in this group will have full access to Deprexis.

INTERVENTIONS:
Behavioral: Deprexis, DeprexisPlus — Online program Deprexis, either as a stand-alone internet-based intervention (Deprexis) or with added standardized email support by a clinical psychologist (DeprexisPlus). In this trial, we will use a Version of Deprexis that has been adapted to MS-specific needs.
  Arms: Deprexis; DeprexisPlus

SUMMARY:
This is an international, multicenter, randomized controlled trial of an internet-based CBT intervention for depression (Deprexis) conducted in five MS centers in the US and Germany. The trial consists of a three-arm primary trial phase and an extension phase targeted at maintenance.

DETAILED DESCRIPTION:
Depression is highly common in MS with a lifetime risk for major depressive disorder (MDD) as high as 25-50% and a 12-month prevalence of up to 25%, particularly in younger patients. Depression in MS has been linked to biological as well as psychological factors and substantially impacts psychosocial function. Importantly, depressive symptoms correlate with decreased quality of life, absence from work, and lower social support and are among the strongest predictors for suicidal ideation in MS patients.

Despite its immediate clinical relevance, depression in MS remains underdiagnosed and often untreated and evidence for the efficacy of pharmacological or non-pharmacological interventions for MS-associated depression is scarce. For example, guidelines recently published by the AAN concluded that evidence for pharmacotherapy and individual or group therapies for MS-depression was insufficient but recommended cognitive behavioral therapy (CBT) delivered by phone with weak level of evidence. Such approaches, however, still require availability of a trained psychotherapist.

Given the mobility problems, cognitive impairment, and fatigue typically associated with MS as well as the limited availability of psychotherapists, self-guided, automated, internet-based interventions may help to overcome treatment barriers often encountered by patients with MS. In a recent phase II randomized controlled trial (RCT) in Germany, the investigators found one such internet-based CBT program, Deprexis, to significantly reduce depressive symptoms in MS (Fischer et al., Lancet Psychiatry 2015). Despite these encouraging results, large, definitive trials of the most promising therapeutic approaches for MS-associated depression that could inform clinical practice are completely lacking.

Here, the investigators conduct a large, international, multicenter RCT of the Deprexis program to treat depression in MS patients. Patients will be recruited in five specialized MS centers in Germany (Charité Berlin and University Medical Center Hamburg) and the US (Cedars Sinai Los Angeles, University of Missouri - Kansas City, and Penn State University). The investigators plan to enroll n=400 patients who will be randomly assigned to two different versions of Deprexis (either Deprexis alone or Deprexis plus regular Email support, DeprexisPlus) for 3 months or a waitlist control group and undergo clinical assessments at baseline and month 3. In addition, the investigators will conduct long-term online follow up at month 6 and month 12.

The trial will address the following three main aims:

Aim 1: To definitively test the effectiveness of Deprexis for reducing depressive symptoms in MS at the end of treatment.

Aim 2: To determine the added value of email support for Deprexis (DeprexisPlus) in MS.

Aim 3: To explore the long-term stability of therapeutic effects (12 months) and the potential of a booster session to enhance maintenance.

ELIGIBILITY:
Inclusion criteria

* age > 18
* neurologist-confirmed diagnosis of MS (all forms)
* self-reported depressive symptoms (BDI-Fastscreen > 4)
* fluent in German or English (depending on study site),
* willingness to engage in self-administration of an iCBT intervention for 3 months and complete follow-up
* ability to travel to the outpatient center for two clinical assessments (baseline and month 3)
* internet access at home

Exclusion criteria:

* unwilling or unable to consent,
* diagnosis of bipolar or psychosis (as determined by M.I.N.I structured interview),
* substantial neurocognitive impairments such as dementia or autism
* moderate or high risk of suicide (according to MINI module C) or by clinical impression
* very severe depression that would interfere with the ability to participate in the study (based on clinical judgment by the physician at the recruitment site).
* current psychotherapy/behavioral treatments for depression
* started pharmacotherapy for depression within the last 2 months
* MS relapse or steroid treatment in the last 4 weeks
* concurrent participation in another clinical trial that includes an intervention
* refusal to saving, processing and forwarding of pseudonymized data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II | Month 0 to Month 3

SECONDARY OUTCOMES:
WHO Quality of Life scale (WHO-QOL BREF) | Month 0 to Month 3
  4 subscales (Physical, Psychological, Social Relationships, Environmental)
Multiple Sclerosis Impact Scale (MSIS) | Month 0 to Month 3
  2 subscales (Physical and Psychological)
Fatigue Scale for Motor and Cognitive Functions (FSMC) | Month 0 to Month 3
  Total score and 2 subscales (Motor and Cognitive)
Chalder Fatigue Scale | Month 0 to Month 3

OTHER OUTCOMES:
Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) | Month 0 to Month 3
  Consists of 3 subtests. 1. SMDT (total score), CVLT-II (2 scores: learning score and delayed recall), and BVMT-R (2 scores: learning score and delayed recall)
Suicide Behaviors Questionnaire-Revised (SBQ-R) | Month 3
Mini International Neuropsychiatric Interview, clinician rating, Version 5.0.0 | Month 0 to Month 3
  Dichotomous variable "Major Depressive Episode, Current (yes/no)" according to module A of the MINI.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Gold, PhD, Study Director — Charité University, Berlin; Friedemann Paul, MD, Principal Investigator — Charité University, Berlin; Christoph Heesen, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Nancy Sicotte, MD, Principal Investigator — Cedars-Sinai Medical Center; Jared Bruce, PhD, Principal Investigator — University of Missouri, Kansas City; Sharon Lynch, MD, Principal Investigator — University of Missouri, Kansas City; Peter Arnett, PhD, Principal Investigator — Penn State University; Rona Moss-Morris, PhD, Principal Investigator — King's College London; Tim Friede, PhD, Principal Investigator — University Medical Center Goettingen; Björn Meyer, PhD, Principal Investigator — GAIA Group
Locations (5):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Missouri, Kansas City, Kansas City, Kansas
  - Penn State University, State College, Pennsylvania
- Germany (2):
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
  - Charité University, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual data on the primary endpoint will be published alongside the trial report in a peer reviewed journal.

REFERENCES:
- [Background] Gold SM, Friede T, Meyer B, Moss-Morris R, Hudson J, Asseyer S, Bellmann-Strobl J, Leisdon A, Issels L, Ritter K, Schymainski D, Pomeroy H, Lynch SG, Cozart JS, Thelen J, Roman CAF, Cadden M, Guty E, Lau S, Pottgen J, Ramien C, Seddiq-Zai S, Kloidt AM, Wieditz J, Penner IK, Paul F, Sicotte NL, Bruce JM, Arnett PA, Heesen C. Internet-delivered cognitive behavioural therapy programme to reduce depressive symptoms in patients with multiple sclerosis: a multicentre, randomised, controlled, phase 3 trial. Lancet Digit Health. 2023 Oct;5(10):e668-e678. doi: 10.1016/S2589-7500(23)00109-7. PMID 37775187